CLINICAL TRIAL: NCT04670484
Title: To Determine the Presence of Mask Hypoxia in Subject Wearing Masks as Personal Protective Equipment (PPE) Due to the Federal Guidelines
Brief Title: Mask Hypoxia in Subjects Using Masks to Prevent Infection Spread
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the cdc and institutional guidelines, study was never started and withdrawn without any enrollment of subjects.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20-456
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2020-12

CONDITIONS: Hypoxia
Keywords: hypoxia; mask
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects wearing masks (Other): Subjects wearing masks to prevent coronavirus infection spread in COVID19 pandemic
  Interventions: Other: Wearing Mask

INTERVENTIONS:
Other: Wearing Mask — Participants wearing masks as per federal guidelines to prevent Coronavirus spread

SUMMARY:
There is some evidence that the use of surgical masks can induce mild hypoxia with a low level of activity (e.g. performing surgery). There is no evidence that this decrease in oxygenation is clinically significant. The degree of hypoxia associated with surgical mask use, N-95 mask use or the combination at rest and with exertion is unclear and warrants further investigation, particularly given the current widespread use of both due to the COVID-19 pandemic. Our working hypothesis is that there is a decrement in oxygenation with the use of any mask that is higher with an N-95 than a surgical mask and higher still when wearing both and that this decrement is more pronounced with exertion than at rest.

DETAILED DESCRIPTION:
Research has shown some evidence of hypoxia associated with the prolonged use of a surgical or N-95 mask. Despite this, the prolonged use of surgical and/or N-95 masks in the clinical setting and surgical masks in the non-clinical setting is the current standard due to the COVID-19 pandemic. The physiologic cost of wearing a respirator was demonstrated in healthy volunteers with mask use during heavy exertion associated with increased respiratory rate, blood pressure and heart rate. N95 use during light exercise increases CO2 intake reduces inspired oxygen and increases the work of breathing. The physiologic effects of N95 fit testing using a hood include higher CO2 levels and lower oxygen levels in the respirator. In patients with ESRD, N95 mask use was associated with reduced PaO2 and increased respiratory rate. The use of surgical masks for prolonged surgeries is associated with decreased SpO2 and increased heart rate, particularly in those over 35 years old. Many studies have suggested that there is a physiologic burden and risk of hypoxia associated with surgical and/or N95 mask use. This pilot study aims to compare baselines with each and both masks and with no mask versus short-duration exertion, which has not yet been done per review of the literature.

There is some evidence that the use of surgical masks can induce mild hypoxia with a low level of activity (e.g. performing surgery) with prolonged use. There is no evidence that this decrease in oxygenation is clinically significant. The degree of hypoxia associated with surgical mask use, N-95 mask use, or the combination at rest and with exertion is unclear and warrants further investigation, particularly given the current widespread use of both due to the COVID-19 pandemic. Our working hypothesis is that there is a decrement in oxygenation with the use of a mask with exertion. The general public is being advised to wear a mask, including those with pre-existing pulmonary disease and heart disease. If there is evidence of a statistically significant decrease in oxygen saturation with short duration mask use with exertion, then further studies on patients at risk for decompensation due to mask-induced hypoxia is warranted. Our working hypothesis is that there is a decrement in oxygenation with the use of a mask with exertion.

This is a single-site study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years old and up wearing masks as personal protective equipment (measure)

Exclusion Criteria:

* Subjects younger than 18 years old.
* Females who are pregnant or women of childbearing potential with a positive pregnancy test at the time of consenting. (If a pregnancy test has not been performed at the time of consenting, the individual will be automatically excluded since a confirmed negative pregnancy test is not available. We will not be able to provide the cost of pregnancy test and will only rely on verbal confirmation from the subject that they are not pregnant or have a -personally purchased standard of care- negative pregnancy test.)
* Consent cannot be obtained from the subject
* Prisoners will be excluded
* Cognitively impaired subjects will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Hypoxia | one year
  Decrease from baseline oxygenation from 70-80% of predicted maximum

IPD SHARING:
Plan to Share IPD: No